CLINICAL TRIAL: NCT01828619
Title: The Study of New RIC Regimen of BuFlu in Older or Intolerable Patients With Hematologic Malignant Diseases
Brief Title: Study of New RIC Regimen of BuFlu in Older and/or Intolerable Patients
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, FENGRONG WANG, Department of Hematology, Peking University People's Hospital
Other Study IDs: PKUIH-201303
Record Dates: First submitted 2013-04-07; First posted 2013-04-10 (Estimated); Last update posted 2013-04-10 (Estimated); Status verified 2013-04

CONDITIONS: Leukemia; Myelodysplastic Syndrome
Keywords: Hematopoietic Stem Cell Transplantation; Busulfan; Fludarabine
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- modified BuFlu, HSCT, elder/intolerable: The study group is the hematlogic malignant patients that older than 55years and/or with severe concurrent medical conditions, who will undergo HLA-matced allogenic HSCT to cure the disease. The patients will received a modified BuFlu conditioning.
  Interventions: Procedure: modified BuFlu conditioning

INTERVENTIONS:
Procedure: modified BuFlu conditioning — The regimen consisted of hydroxyurea 80 mg/kg on d -10; cytorabine 2 g/m2 on d -9; busulfan 3.2mg/kg/day iv. ×3days( on d -8 to -6); Flu30mg/m^2 i.v.×5days(on d-6 to-2) and semustine 250 mg/m2 on d -3.

SUMMARY:
The purpose of this study is to determine whether the new RIC regimen, containing of low dose of Bu (9.6mg/kg)and fludarabine without ATG, is suitable and effective in treating aged and/or intolerable patients with hematologic malignant disease, who undergoes allogenic stem cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed of hematologic malignant disease
* will undergo HLA matced HSCT
* age >=55years
* <55year and intolerable to standard myeloablative conditioning

Exclusion Criteria:

* KPS status <70
* cardiac EF<50%
* creatine clearance <50 ml/min
* ALT more than 10 times of upper normal limit

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is patients with hematologic malignant diseases, who will undergo HLA matched HSCT.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2013-02; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
stem cell engraftment | 30day post transplantation

SECONDARY OUTCOMES:
toxicity and treatment related mortality | 100day and 1 year post transplantation

CONTACTS AND LOCATIONS:
Overall Officials: XiaoJun Huang, MD, Principal Investigator — Peking University People's Hospital, Department of Hematology
Locations (1):
- Peking University People's Hospital, Beijing, China

REFERENCES:
- [Background] Barrett AJ, Savani BN. Stem cell transplantation with reduced-intensity conditioning regimens: a review of ten years experience with new transplant concepts and new therapeutic agents. Leukemia. 2006 Oct;20(10):1661-72. doi: 10.1038/sj.leu.2404334. Epub 2006 Jul 27. PMID 16871277
- [Background] de Lima M, Couriel D, Thall PF, Wang X, Madden T, Jones R, Shpall EJ, Shahjahan M, Pierre B, Giralt S, Korbling M, Russell JA, Champlin RE, Andersson BS. Once-daily intravenous busulfan and fludarabine: clinical and pharmacokinetic results of a myeloablative, reduced-toxicity conditioning regimen for allogeneic stem cell transplantation in AML and MDS. Blood. 2004 Aug 1;104(3):857-64. doi: 10.1182/blood-2004-02-0414. Epub 2004 Apr 8. PMID 15073038